CLINICAL TRIAL: NCT06856824
Title: Functional Results of Infiltration for Biceps Tendonitis Guided by Ultrasound vs Anatomical Repairs: Variation in Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024/070
Record Dates: First submitted 2024-05-16; First posted 2025-03-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Bíceps Tendinitis
Keywords: Bíceps; Tendinitis; injection; ultrasound; corticosteroid
MeSH Terms: conditions — Tendinopathy | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anatomic landmarks (Active Comparator): injection in the bicipital groove guided by anatomic landmarks
  Interventions: Procedure: injection in the bicipital groove guided by anatomic landmarks
- Guided by ultrasound (Experimental): injection in the bicipital groove guided by ultrasound
  Interventions: Procedure: injection in the bicipital groove guided by ultrasound

INTERVENTIONS:
Procedure: injection in the bicipital groove guided by anatomic landmarks — Anatomical landmark-guided puncture involves patient positioning and palpation, whereas ultrasound-guided involves identifying the biceps tendon's axis and inserting the needle parallel to the transducer.
  Arms: Anatomic landmarks
Procedure: injection in the bicipital groove guided by ultrasound — Anatomical landmark-guided puncture involves patient positioning and palpation, whereas ultrasound-guided involves identifying the biceps tendon's axis and inserting the needle parallel to the transducer.
  Arms: Guided by ultrasound

SUMMARY:
A randomized clinical trial aimed at comparing the functional outcomes of brachial biceps infiltration guided by anatomical landmarks versus ultrasound guidance. Given that ultrasound guidance has shown an efficacy of 91%, this intervention could potentially be more effective in delivering medication to the target area and achieving improved therapeutic outcomes

DETAILED DESCRIPTION:
Shoulder pain is a frequent orthopedic complaint, with biceps long head tendinitis being a common cause leading to physical disability in the working and athletic population. Currently, there's no guideline for managing biceps tendinitis. Studying clinical outcomes post-biceps tendon sheath infiltration will aid in developing management guidelines for quick patient return to activities with minimal sequelae.

No studies in Colombia have compared clinical outcomes of biceps tendinitis patients undergoing ultrasound-guided vs anatomically guided infiltrations. This information will allow comparison with global literature, assessing differences in treatment effectiveness and socio-economic impact on the population.

Research Question:

In patients with long head biceps tendinitis, does ultrasound-guided infiltration compared to anatomically guided infiltration yield better clinical outcomes?

Theoretical Framework and State of the Art:

The biceps tendon originates from the supraglenoid tubercle of the scapula, contributing to shoulder stability and functions such as forearm supination and elbow flexion. Primary biceps tendinitis, constituting about 5% of bicipital pathology cases, can limit daily activities.

Tendinitis cascade initiation involves inflammation due to repetitive traction, leading to increased tendon volume and pressure in specific locations, predisposing it to shear forces and degenerative changes. Diagnosis involves ultrasound and MRI, with initial treatment focusing on non-surgical methods and corticosteroid infiltrations when conservative management fails.

Ultrasound-guided injections, compared to anatomical landmarks, show higher precision and efficacy rates, reducing patient discomfort.

Procedure Technique:

Anatomical landmark-guided puncture involves patient positioning and palpation, whereas ultrasound-guided involves identifying the biceps tendon's axis and inserting the needle parallel to the transducer.

Objectives:

General Objective: To compare functional outcomes of biceps tendon sheath infiltration guided by anatomical landmarks versus ultrasound in biceps tendinitis patients.

Specific Objectives: Characterize patient demographics, describe complication incidence, compare complication incidence between groups, and compare clinical outcomes between techniques.

Hypotheses:

Null Hypothesis: Ultrasound-guided infiltration yields similar functional results as anatomical landmark-guided infiltration in biceps tendinitis patients.

Alternative Hypothesis: Ultrasound-guided infiltration yields better functional results than anatomical landmark-guided infiltration in biceps tendinitis patients.

Methodology:

This entails a randomized clinical trial with double-blind methodology, involving RedCap software for randomization. Patients are blinded to the procedure, while the applicator knows the procedure but outcome evaluators are blinded.

Anatomical Landmark-guided Puncture:

The patient is placed in the supine position with the shoulder at a 10° internal rotation angle. Identification involves palpation of the coracoid process, tuberosities, biceps tendon, and bicipital groove. The tuberosities and biceps tendon groove are marked at the presumed tendon location. Confirmation of tendon location is achieved through palpation with rotations and manual palpation (highlighting 5 to 7 cm distal to the anterolateral margin of the acromion). A 5cc syringe with a 0.8 x 40 mm 21G ½ needle is used for puncture, inclined at a 20° to 30° cephalic angle until the biceps tendon sheath is pierced. During the procedure, ultrasound machine and transducer positioning will be performed, although the device will remain turned off.

Ultrasound-guided Puncture:

The patient is positioned supine with the shoulder in a neutral rotation. Identification involves locating the axis of the long head biceps tendon. The transducer is positioned perpendicular to the synovial sheath. The needle is inserted parallel to the transducer along its long axis from the lateral side of the shoulder. The needle is visualized on the monitor as a hyperechoic image and advanced continuously and in real-time into the tendon sheath. A 5cc syringe with a 0.8 x 40 mm 21G ½ needle is used for puncture. This procedure is performed by a specialist trained in ultrasound.

General Objective Compare the functional outcomes of bicipital groove infiltration guided by anatomical landmarks and by ultrasound as a technique variation in patients with biceps tendinitis.

Specific Objectives

Characterize demographic variables in the study patient groups. Describe the incidence of complications related to the procedures. Compare the incidence of complications between the groups. Compare clinical outcomes between the two techniques (EVA, qDASH, SANE, satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients with anterior shoulder pain
* Point of maximum pain in long head bíceps tendon at the level of the bicipital groove
* Positive speed test
* Patients who gave informed consent and accepted follow-up

Exclusion Criteria:

* Calcifying tendonitis of the biceps
* Partial or complete rupture of the subscapularis tendon
* Glenohumeral joint deformity
* Rupture and/or dislocation of the tendon of the long head of the biceps.
* Surgery and/or previous infiltrations in the biceps tendon

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
qDASH | initial measurement before treatment administration, final measurement at 4 weeks.
  The QuickDASH, published in 2005 in the Journal of Bone and Joint Surgery, is an 11-item subset of the 30-item DASH and is a self-report questionnaire in which response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and scores range from MINIMUM 0 to 100. 0 is the minimum score and 100 is the maximum score. 0 indicates no disability and 100 indicates more severe disability. Higher scores indicate worse outcome. This score was designed to be useful in patients with any upper extremity musculoskeletal disorder.
SANE | initial measurement before treatment administration, follow up at 1, 2, 3 and 4 months
  The Single Assessment Numeric Evaluation (SANE) is a quick assessment tool that asks patients to rate their affected joint function as a percentage of normal, where 100% represents normal function and 0% indicates completely abnormal function.
  Thus, the maximum score is 100%, and the minimum is 0%. A higher score reflects a better perception of function by the patient. For example, a score of 85% suggests that the patient perceives their joint function at 85% of what they consider normal.
  Studies have shown that initial SANE scores typically range between 40% and 60% before treatment, improving to 75% to 85% one year after therapy, depending on the condition treated.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) for Pain Assessment | initial measurement before treatment administration, follow up at 1, 2, 3 and 4 months
  The VAS is a widely used unidimensional tool for assessing pain intensity in clinical and research settings. It consists of a 10 cm horizontal line where one end represents "no pain" (0 cm) and the other "the worst pain imaginable" (10 cm). The patient is asked to place a mark on the line corresponding to their perceived pain level, and the score is determined by measuring the distance from the "no pain" anchor to the patient's mark in centimeters.
  Assessment Method:
  Patients self-report pain by marking a continuous 10 cm line. Pain intensity is quantified by measuring the mark's distance in millimeters (mm) from the zero point (0 mm = no pain, 100 mm = worst pain imaginable).
  Interpretation:
  0-4 mm: No pain 5-44 mm: Mild pain 45-74 mm: Moderate pain 75-100 mm: Severe pain
Tenderness to palpation | Time Frame initial measurement before treatment administration, final measurement at 4 months.
  Pain or discomfort at palpation in the bicipital groove, the escale use is VAS por sus siglas en inglés: Visual Analogue Scale. It consists of a horizontal line of 10 cm (or 100 mm), where one end represents "no pain" (0) and the other end "the worst pain imaginable" (10 or 100, depending on the scale used). The higher the scale value, the worse the patient's health condition and the greater the pain.
Speed Test | Time Frame initial measurement before treatment administration, final measurement at 4 months.
  the patient is asked to extend his elbow and fully supinate his forearm again and to bring his shoulder into 90 degrees of flexion. In this position, the patient is asked to resist downward pressure.the biceps tendon acts like a suspensor cable from its insertion on the superior labrum to the arm. Increased tension in this cable and if inflammation is present is thought to result in pain in the proximal shoulder
Yergason Test | initial measurement before treatment administration, final measurement at 4 months.
  The patient should be seated or standing in the anatomical position, with the humerus in a neutral position and the elbow in 90 degrees of flexion in a pronated position. The patient is asked to externally rotate and supinate their arm against the manual resistance of the therapist produced by wrapping the hand around the distal forearm (just above the wrist joint).[2] Yergason's Test is considered positive if the pain is reproduced in the bicipital groove and a biceps or a SLAP lesion is suspected. If a "clicking" sensation familiar to the patient is produced during the test, damage to the transverse humeral ligament (which overlies the intertubercular sulcus) should be suspected too
Satisfaction with treatment | final measurement at 4 months.
  Satisfaction with treatment is a patient-reported outcome that assesses the perceived effectiveness of the intervention in terms of pain relief and functional recovery.
  Measurement Tool:
  Question Format: Binary (Yes/No) Type of Variable: Quantitative (Dichotomous)
  Assessment Method: Patients will be directly asked:
  "Are you satisfied with the treatment in terms of pain relief and functional recovery?" Yes (1): The patient reports being satisfied. No (0): The patient reports not being satisfied.
  Interpretation:
  A higher percentage of "Yes" responses indicates a greater overall treatment satisfaction rate.
Complications | final measurement at 4 months.
  patients will be evaluated in terms of infection development and biceps tendon rupture as principal complications

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aly AR, Rajasekaran S, Ashworth N. Ultrasound-guided shoulder girdle injections are more accurate and more effective than landmark-guided injections: a systematic review and meta-analysis. Br J Sports Med. 2015 Aug;49(16):1042-9. doi: 10.1136/bjsports-2014-093573. Epub 2014 Nov 17. PMID 25403682
- [Result] Urwin M, Symmons D, Allison T, Brammah T, Busby H, Roxby M, Simmons A, Williams G. Estimating the burden of musculoskeletal disorders in the community: the comparative prevalence of symptoms at different anatomical sites, and the relation to social deprivation. Ann Rheum Dis. 1998 Nov;57(11):649-55. doi: 10.1136/ard.57.11.649. PMID 9924205
- [Result] Holtby R, Razmjou H. Accuracy of the Speed's and Yergason's tests in detecting biceps pathology and SLAP lesions: comparison with arthroscopic findings. Arthroscopy. 2004 Mar;20(3):231-6. doi: 10.1016/j.arthro.2004.01.008. PMID 15007311
- [Result] Dean BJ, Gwilym SE, Carr AJ. Why does my shoulder hurt? A review of the neuroanatomical and biochemical basis of shoulder pain. Br J Sports Med. 2013 Nov;47(17):1095-104. doi: 10.1136/bjsports-2012-091492. Epub 2013 Feb 21. PMID 23429268
- [Result] Borms D, Ackerman I, Smets P, Van den Berge G, Cools AM. Biceps Disorder Rehabilitation for the Athlete: A Continuum of Moderate- to High-Load Exercises. Am J Sports Med. 2017 Mar;45(3):642-650. doi: 10.1177/0363546516674190. Epub 2016 Dec 14. PMID 28125910
- [Result] Griffin JW, Leroux TS, Romeo AA. Management of Proximal Biceps Pathology in Overhead Athletes: What Is the Role of Biceps Tenodesis? Am J Orthop (Belle Mead NJ). 2017 Jan/Feb;46(1):E71-E78. PMID 28235123
- [Result] Varacallo MA, Mair SD. Proximal Biceps Tendinitis and Tendinopathy. 2023 Aug 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK533002/ PMID 30422594
- [Result] Arroll B, Goodyear-Smith F. Corticosteroid injections for painful shoulder: a meta-analysis. Br J Gen Pract. 2005 Mar;55(512):224-8. PMID 15808040
- [Result] Buchbinder R, Green S, Youd JM. Corticosteroid injections for shoulder pain. Cochrane Database Syst Rev. 2003;2003(1):CD004016. doi: 10.1002/14651858.CD004016. PMID 12535501
- [Result] Zhang J, Ebraheim N, Lause GE. Ultrasound-guided injection for the biceps brachii tendinitis: results and experience. Ultrasound Med Biol. 2011 May;37(5):729-33. doi: 10.1016/j.ultrasmedbio.2011.02.014. Epub 2011 Mar 31. PMID 21458143
- [Result] Elkousy H, Gartsman GM, Drake G, Sola W Jr, O'Connor D, Edwards TB. Retrospective comparison of freehand and ultrasound-guided shoulder steroid injections. Orthopedics. 2011 Apr 11;34(4). doi: 10.3928/01477447-20110228-11. PMID 21469629
- [Result] González FSV, Shoji FH, Díaz MIE. Lesiones del tendón del bíceps, manejo actual. Orthotips AMOT 2014;10:154-62.
- [Result] Khazzam M, George MS, Churchill RS, Kuhn JE. Disorders of the long head of biceps tendon. J Shoulder Elbow Surg. 2012 Jan;21(1):136-45. doi: 10.1016/j.jse.2011.07.016. Epub 2011 Oct 17. No abstract available. PMID 22005126
- [Result] García González GLA, Aguilar Sierra SF, Rodríguez Ricardo RMC. Validación de la versión en español de la escala de función del miembro superior abreviada: Quick Dash. Revista Colombiana de Ortopedia Y Traumatología 2018;32:215-9.
- [Result] Dhand NK, Khatkar MS. Statulator: An online statistical calculator. Sample size calculator for comparing two independent means. Accessed May 2014;6:2021.